CLINICAL TRIAL: NCT06038799
Title: Caregiver Skills Training: Comparing the Effectiveness of Training Clinicians Via Telehealth and In-Person Training
Brief Title: Caregiver Skills Training: Comparing Clinician Training Methods
Acronym: CST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: poor subject accrual; unable to meet study aims
Sponsor: University of Pittsburgh (Other)
Collaborators: Autism Speaks (Other)
Responsible Party: Principal Investigator, Benjamin L Handen, PhD, BCBA-D, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY23040076
Record Dates: First submitted 2023-07-19; First posted 2023-09-15 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Parenting
Keywords: Caregiver skills training; Staff training

STUDY DESIGN:
Intervention Model Description: The investigators will be comparing two types of training/supervision models. One will be provided remotely and one will be provided face-to-face. In addition, investigators will compare two types of treatment: face-to-face sessions versus remote sessions.
Who Masked: Care Provider
Masking Description: Parents that receive Caregiver Skills Training will be unaware of whether their group leaders were trained/supervised remotely or face-to-face.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remote staff training (Active Comparator): Staff will receive 15 hours of remote training followed by 12 weeks of remote supervision (one hour per week).
  Interventions: Behavioral: Caregiver Skills Training (CST)
- Face to face staff training (Active Comparator): Staff will receive 15 hours of face to face training followed by 12 weeks of face to face supervision (one hour per week).
  Interventions: Behavioral: Caregiver Skills Training (CST)

INTERVENTIONS:
Behavioral: Caregiver Skills Training (CST) — The investigators are comparing the relative efficacy of CST between a CST group led by clinicians trained and supervised remotely versus a group led by clinicians trained an supervised face-to-face.

SUMMARY:
Caregiver Skills Training (CST) is an evidence-based intervention for parents of young children with developmental disabilities that was developed through a collaboration between Autism Speaks and the World Health Organization. The intervention is typically offered by Facilitators who are trained and supervised by CST Master Trainers. This study seeks to use a remote training model to compare two training and supervision processes. One group, comprised of facilitators from rural settings, will be trained and supervised by two master trainers from the University of Pittsburgh using a remote training model. A second group, comprised of facilitators from an agency serving primarily low-income households and located near Pittsburgh, will be trained and supervised in a face-to-face manner. Both groups will initially receive ten 90-minute training sessions over a 2-month period and will subsequently receive 1 hour per week of supervision while conducting their first 12-session CST group. Outcome measures will include assessment of change in caregiver stress and didactic skills as well as improvement in each child's communication/social skills, functional skills, and overall behavior. Also added was an additional research question in which face-to-face CST sessions with remote CST sessions were compared.

DETAILED DESCRIPTION:
There are two aspects to this study: First, the investigators will compare two training and supervision processes. One group, comprised of facilitators from rural settings, will be trained and supervised by two master trainers from the University of Pittsburgh Medical Center (UPMC) Center for Autism and Developmental Disorders (CADD). A second group, comprised of facilitators from an agency serving primarily low-income households and located near Pittsburgh, PA, will be trained and supervised in a face-to-face manner. Both groups will receive 15 hours of training spread over the course of 2-3 months (in summer 2023). The focus of these sessions will be to introduce and train staff on the CST model, ensure their understanding of the curriculum, and to help them gain proficiency in administration. During the training phase, both groups will practice administration of activities and will be provided feedback. The master trainers will also assist the newly trained facilitators in navigating recruitment and organization of their first CST groups. Upon initiation of the CST groups, facilitators will receive 1 hour of supervision per week, either in person or via TEAMS. Supervision will extend over the 9 group sessions and 3 home visits per family (fall 2023). These supervision sessions will allow the facilitators to ask questions, obtain feedback, and troubleshoot any challenges. The investigators will also collect pre and post measures (baseline and week 12) from the parents participating in the CST groups to determine if the type of training provided to the facilitators (face-to-face versus remote) impacted parent progress. We have also added an additional research question in which we compare face-to-face CST sessions with remote CST sessions.

ELIGIBILITY:
Inclusion Criteria:

Parents who

* Have a child ages 2-9 with a developmental disability and/or autism
* Able to be served by one of the three UPMC sites
* Able to attend 12 sessions. Group sessions are at the clinic site and the individual sessions may be done virtually or in person.

Exclusion Criteria:

* Parent()s does not speak / understand English. Given the nature of this study, we are unable to provide translation services.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change from week 1 (baseline) to week 12 on the Caregivers Skills and Knowledge Measure | Week 1 (baseline) versus week 12 (final visit)
  eEvaluates change in caregiver skills and knowledge related to session content as well as caregiver confidence. There are 28 skills questions (scored on a scale of 1-5) with a score range fomr 28-140 (with higher scores indicating greater skills). The Confidence scale consists of 9 items (scored 1-5) with scores ranging from 9-45. Higher scores indicate greater confidence.

SECONDARY OUTCOMES:
Change from week 1 (baseline) to week 12 on the Parenting Stress Index. | Week 1 (baseline) versus week 12 (final visit)
  To assess parental distress, parent-child dysfunctional interaction, and child challenges. There are 36 items and 3 subscales (12 items per subscale). Subscales include Parent Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. There is also a Total Stress Score. Each item is scored on a 1-5 scale. Range for each subscale is 12-60 points; Total Score is 36-180 points. Scores are converted to percentiles. Percentiles of 15-80 are "typical stress;" 81-89 are "high stress;" and >89 are "clinically significant stress." Higher percentiles indicate higher levels of stress.
Change from week 1 (baseline) to week 12 on the Social Communication Checklist (SCC) | Week 1 (baseline) versus week 12 (final visit)
  To assess social communication abilities, specifically social engagement (15 items), expressive language form (15 items), expressive language function (15 items), receptive language (8 items) imitation (6 items, and pla (11 items). Items are scored on a 3-point scale ("usually," = 3 points; "sometimes," = 2 points; or "rarely" = 1 point). The range for all 70 items is 70-210 points. The higher the score, the greater the child's abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Handen, PhD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC Mon Yough, McKeesport, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the study protocol, consent, analysis plan and results upon request by qualified researchers/professionals.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The study protocol, consent form, and statistical analysis plan are available now (as of 9/8/23).The investigators hope to complete the data analysis by late spring 2024 (within 1 year of study completion) and will make a CSR available at that time.
Access Criteria: Interested investigators should contact the PI directly, who will review requests.

REFERENCES:
- [Background] Ludwig NN, Suskauer SJ, Rodgin S, Chen J, Borda A, Jones K, Lahey S, Slomine BS. Outcome Measurement in Children With a History of Disorders of Consciousness After Severe Brain Injury: Telephone Administration of the Vineland Adaptive Behavior Scales, Third Edition, and Glasgow Outcome Scale-Extended Pediatric Revision. Pediatr Crit Care Med. 2023 Feb 1;24(2):e76-e83. doi: 10.1097/PCC.0000000000003121. Epub 2022 Dec 16. PMID 36661427
- [Background] Holly LE, Fenley AR, Kritikos TK, Merson RA, Abidin RR, Langer DA. Evidence-Base Update for Parenting Stress Measures in Clinical Samples. J Clin Child Adolesc Psychol. 2019 Sep-Oct;48(5):685-705. doi: 10.1080/15374416.2019.1639515. Epub 2019 Aug 8. PMID 31393178
- [Background] Wainer AL, Berger NI, Ingersoll BR. Brief Report: The Preliminary Psychometric Properties of the Social Communication Checklist. J Autism Dev Disord. 2017 Apr;47(4):1231-1238. doi: 10.1007/s10803-016-3026-8. PMID 28105548
- [Background] Sengupta K, Shah H, Ghosh S, Sanghvi D, Mahadik S, Dani A, Deshmukh O, Pacione L, Dixon P, Salomone E; WHO-CST team; Servili C. World Health Organisation-Caregiver Skills Training (WHO-CST) Program: Feasibility of Delivery by Non-Specialist Providers in Real-world Urban Settings in India. J Autism Dev Disord. 2023 Apr;53(4):1444-1461. doi: 10.1007/s10803-021-05367-0. Epub 2021 Dec 1. PMID 34853959
- [Background] Kasari C, Lawton K, Shih W, Barker TV, Landa R, Lord C, Orlich F, King B, Wetherby A, Senturk D. Caregiver-mediated intervention for low-resourced preschoolers with autism: an RCT. Pediatrics. 2014 Jul;134(1):e72-9. doi: 10.1542/peds.2013-3229. PMID 24958585